CLINICAL TRIAL: NCT02387710
Title: Inducing Slow Wave Sleep to Treat Obstructive Sleep Apnea
Brief Title: Tiagabine to Enhance Slow Wave Sleep in Patients With Sleep Apnea
Acronym: TESSA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, David Andrew Wellman, Director, Sleep Disordered Breathing Laboratory, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BWH-2012P000956B
Record Dates: First submitted 2015-03-09; First posted 2015-03-13 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2017-07

CONDITIONS: Sleep Apnea, Obstructive
Keywords: arousal threshold; phenotype; tiagabine; slow wave sleep
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Tiagabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tiagabine (Active Comparator): Tiagabine PO 12 mg before sleep
  Interventions: Drug: Tiagabine
- Placebo (Placebo Comparator): Placebo PO before sleep
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tiagabine — GABA reuptake inhibitor
  Other Names: Gabitril
  Arms: Tiagabine
Drug: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
Obstructive sleep apnea (OSA) is common and has major health implications but treatment options are limited. Interestingly, the severity of OSA is profoundly reduced in deep sleep (called "slow wave sleep"), potentially via an increase in the stimulus required to arouse from sleep. Here the investigators test the idea that the medication called "tiagabine" improves slow wave sleep and reduces OSA severity. The investigators will also test whether tiagabine raises the arousal threshold (more negative esophageal pressure), and whether detailed OSA "phenotyping" characteristics can predict the improvement in OSA severity with this intervention.

DETAILED DESCRIPTION:
The current study tests the primary hypothesis that tiagabine improves sleep apnea severity in patients with moderate-to-severe sleep apnea (apnea hypopnea index measured in supine non-REM sleep; hypopneas defined by 3% desaturation or arousal). The investigators test three secondary hypotheses that tiagabine:

1. increases the proportion of total sleep time in slow wave sleep
2. raises the non-REM arousal threshold (more negative esophageal pressure) via (1).
3. is preferentially effective in patients whose OSA phenotype predicts that an increase in the arousal threshold is sufficient to resolve OSA versus those without such favorable physiology. Favorable physiology is defined here as having a low ventilatory drive at which stable breathing is theoretically feasible ("stable Vdrive" is <100% above eupneic ventilatory drive) due to any combination of a "high" upper airway muscle response, "good" passive anatomy (high Vpassive), and "low" steady-state loop gain (see Owens RL et al SLEEP 2014; Wellman A et al J Appl Physiol 2011, 2013; Eckert DJ et al 2013 AJRCCM).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed OSA (moderate-to-severe; apnea hypopnea index >15 events/hr)

Exclusion Criteria:

* History of seizures

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-03; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sleep Disorders Research Program Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Taranto-Montemurro L, Sands SA, Edwards BA, Azarbarzin A, Marques M, de Melo C, Eckert DJ, White DP, Wellman A. Effects of Tiagabine on Slow Wave Sleep and Arousal Threshold in Patients With Obstructive Sleep Apnea. Sleep. 2017 Feb 1;40(2):zsw047. doi: 10.1093/sleep/zsw047. PMID 28364504

RESULTS

PARTICIPANT FLOW:
Groups:
- Tiagabine First, Placebo Second: Tiagabine 12 mg administered at normal sleep time on first study night, then a 1-week non-treatment period, then placebo-matching tiagabine administered at normal sleep time on second study night.
- Placebo First, Tiagabine Second: Placebo-matching tiagabine administered at normal sleep timeon first study night, then a 1-week non-treatment, then tiagabine 12 mg administered at normal sleep time on second study night
Period: First Study Night
Arm/Group | Tiagabine First, Placebo Second | Placebo First, Tiagabine Second
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0
Period: Second Study Night
Arm/Group | Tiagabine First, Placebo Second | Placebo First, Tiagabine Second
Started | 9 | 7 (2 patients did not come back for excessive sleep disruption due to the equipment)
Completed | 9 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 18 patients enrolled, 2 did not completed the study, One patient was excluded because of predominantly central sleep apnea on both nights, and another was excluded because of low-quality EEG data. Therefore, 14 subjects were analyzed.
Groups:
- All Analyzed Participants: All patients who were randomized, completed both study nights and were included in the analysis
Arm/Group | All Analyzed Participants
Number analyzed (Participants) | 14
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [51 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Apnea Hypopnea Index (AHI)
Description: Number of apneas + hypopneas per hour of sleep. Hypopnea criteria: reduction in 30% of baseline flow plus 3% desaturation or arousal.
Time Frame: 1 night
Measure: Median (Inter-Quartile Range); unit: events/hour
Groups:
- Tiagabine: Tiagabine 12 mg administered at sleep time on the first or second study night
- Placebo: Placebo administered at sleep time on the first or second study night
Arm/Group | Tiagabine | Placebo
Number analyzed (Participants) | 14 | 14
events/hour | 39.1 [32.1 to 48.7] | 40.8 [31.4 to 51.7]
Statistical Analysis 1: Comparison: Tiagabine vs Placebo; Test type: Other; p > 0.5, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Slow Wave Sleep (% Total Sleep Time)
Description: Fraction of sleep spent in stage N3
Time Frame: 1 night
Measure: Median (Inter-Quartile Range); unit: % total sleep time
Arm/Group | Tiagabine | Placebo
Number analyzed (Participants) | 14 | 14
% total sleep time | 8.3 [4.52 to 20.6] | 8.8 [5.2 to 15.7]

3. Secondary Outcome: Arousal Threshold (Esophageal Pressure Swing)
Description: The arousal threshold was quantified as the mean of all the nadir negative esophageal pressure swings immediately preceding an arousal at the end of an obstructive apnea or hypopnea during both placebo and tiagabine nights.
Time Frame: 1 night
Measure: Median (Inter-Quartile Range); unit: cmH2O
Groups:
- Tiagabine: Tiagabine 12 mg administered at sleep time on the first or the second study night
- Placebo: Placebo administered at sleep time on the first or the second study night
Arm/Group | Tiagabine | Placebo
Number analyzed (Participants) | 14 | 14
cmH2O | -27.6 [-28.6 to -23.6] | -26.5 [-27.9 to -23]

ADVERSE EVENTS:
Arm/Group | Tiagabine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes